CLINICAL TRIAL: NCT04679948
Title: The Effect of Multiple Doses of BI 730357 on the Single Dose Pharmacokinetics of Caffeine, Warfarin, Omeprazole and Midazolam Administered Orally as a Cocktail in Healthy Subjects (an Open-label, Two-period Fixed Sequence Design Trial)
Brief Title: A Study in Healthy People to Test Whether BI 730357 Influences the Amount of Caffeine, Warfarin, Omeprazole, and Midazolam in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1407-0039; 2020-002506-51 (EudraCT Number)
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Healthy
MeSH Terms: interventions — Caffeine; Warfarin; Omeprazole; Midazolam

STUDY DESIGN:
Intervention Model Description: Two Periods (Period 1 and Period 2) for each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cocktail/ Cocktail + BI 730357 (Experimental): Cocktail treatment will be followed by the Test treatment (Cocktail + BI 730357) in a fixed sequence. The treatment periods are separated by a wash-out phase of at least 20 days between the two cocktail administrations.
  Interventions: Drug: Percoffedrinol®; Drug: Coumadin®; Drug: Antra MUPS®; Drug: Midazolam-ratiopharm®; Drug: BI 730357

INTERVENTIONS:
Drug: Percoffedrinol® — Tablet
  Other Names: Caffeine
Drug: Coumadin® — Tablet
  Other Names: Warfarin sodium
Drug: Antra MUPS® — Gastro-resistant tablet
  Other Names: Omeprazole
Drug: Midazolam-ratiopharm® — Oral solution
  Other Names: Midazolam
Drug: BI 730357 — Film-coated tablet

SUMMARY:
The trial will be performed to assess the influence of BI 730357 on the pharmacokinetics of caffeine, warfarin, omeprazole and midazolam.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation
* Either male subject, or female subject who meet any of the following criteria from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Use of non-hormonal intrauterine device plus condom for birth control
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
  * Surgically sterilised (including hysterectomy or bilateral tubal occlusion)
  * Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with levels of follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR, or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract (except appendectomy or simple hernia repair) that could interfere with the pharmacokinetics (PK) of the trial medication
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further inclusion exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase 1, non-randomised, open-label, 2-treatment, 2-period fixed sequence design trial in healthy people to test whether BI 730357 influences the amount of caffeine, warfarin, omeprazole, and midazolam in the blood.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Drug Cocktail Alone (R) Then Drug Cocktail + BI 730357 (T): In period 1: Participants were administered the cocktail reference treatment (R) consisting of 2 tablets of 50 milligrams (mg) (total dose 100mg) of caffeine (Percoffedrinol® N 50 mg Tablets), 2 tablets of 5 mg (total dose 10 mg) of warfarin sodium (Coumadin® 5 mg), 1 tablet of 20 mg of omeprazole (Antra MUPS® 20 mg gastro-resistant tablet), and 1 milliliter (mL) oral solution of 2 mg of midazolam (Midazolam-ratiopharm® 2 mg/mL oral solution), each medication as a single dose, once on Day 1 of period 1 (Visit 2).
  In period 2 (Visit 3): Participants were administered 3 film-coated tablets of 100 mg BI 730357 orally twice daily (bid) (daily dose 600 mg) from Day -14 to Day 6 of Visit 3 (20 days in total). On the 15th day of BI 730357 treatment (Day 1 of Visit 3, 1 h after the morning dose of BI 730357), the cocktail (100 mg caffeine, 10 mg warfarin, 20 mg omeprazole, and 2 mg midazolam) was administered orally once. The BI 730357+ cocktail was the test treatment (T).
  The two cocktail administrations were separated by a wash-out period of at least 20 days.
Period: Period 1
Arm/Group | Drug Cocktail Alone (R) Then Drug Cocktail + BI 730357 (T)
Started | 16
Completed | 16
Not Completed | 0
Period: Period 2
Arm/Group | Drug Cocktail Alone (R) Then Drug Cocktail + BI 730357 (T)
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all subjects who were entered and treated with at least 1 dose of trial drug.
Arm/Group | Drug Cocktail Alone (R) Then Drug Cocktail + BI 730357 (T)
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Caffeine in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity, Caffeine)
Description: Area under the concentration-time curve of caffeine in plasma over the time interval from 0 extrapolated to infinity (AUC0-infinity, caffeine) is reported.
Time Frame: Within 2 hours (h) predose for period 1, within 15 minutes predose for period 2 and 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 48 h after caffeine administration in both periods.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This set included all subjects in the TS who provided at least 1 PK endpoint that was defined as primary and was not excluded due to a clinical trial protocol (CTP) deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS, even if the subject contributed only 1 PK parameter value for 1 period to the statistical assessment. Only those with non-missing results are included in the analysis.
Measure: Geometric Least Squares Mean (Standard Error); unit: hours *nanomole/Liter (h*nmol/L)
Groups:
- Caffeine (Reference (R)): In period 1 (Visit 2): Participants were administered 2 tablets of 50 milligrams (mg) (total dose 100 mg) of caffeine (Percoffedrinol® N 50 mg tablets) orally as a single dose once on Day 1 of period 1 (Visit 2).
- BI 730357 + Caffeine (Test (T)): In period 2 (Visit 3): Participants were administered 3 film-coated tablets of 100 mg BI 730357 orally twice daily (bid) with daily dose 600 mg from Day -14 to Day 6 of Visit 3 (20 days in total). On the 15th day of BI 730357 treatment (Day 1 of Visit 3, 1 h after the morning dose of BI 730357), 2 tablets of 50 milligrams (mg) (total dose 100 mg) of caffeine (Percoffedrinol® N 50 mg tablets) were administered orally once. The two caffeine administrations were separated by a wash-out period of at least 20 days.
Arm/Group | Caffeine (Reference (R)) | BI 730357 + Caffeine (Test (T))
Number analyzed (Participants) | 15 | 15
hours *nanomole/Liter (h*nmol/L) | 84569.29 (NA) — Adjusted geometric standard error=1.11 | 94764.64 (NA) — Adjusted geometric standard error=1.11
Statistical Analysis 1: Comparison: Caffeine (Reference (R)) vs BI 730357 + Caffeine (Test (T)); The statistical model used for the analysis of the primary endpoints was an analysis of variance (ANOVA) model on the logarithmic scale. That is, the PK endpoints were logtransformed (natural logarithm) prior to fitting the ANOVA model. These quantities were then back-transformed to the original scale to provide the point estimate and 90% CIs for each endpoint. This model included effects accounting for the following sources of variation: subjects (random effect) and treatment (fixed effect); Test type: Other; Ratio of GLSMs [%] = 112.06, 90% CI 2-sided [101.02 to 124.30] — Ratio of Geometric Least Squares Means (GLSMs) was calculated as (GLSM of "BI 730357 + caffeine"/GLSM of "caffeine"). Intra-individual geometric coefficient of variation (gCV [%]) =16.2

2. Primary Outcome: Maximum Measured Concentration of the Caffeine in Plasma (Cmax, Caffeine)
Description: Maximum measured concentration of the caffeine in plasma (Cmax, caffeine) is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/Liter (nmol/L)
Arm/Group | Caffeine (Reference (R)) | BI 730357 + Caffeine (Test (T))
Number analyzed (Participants) | 15 | 15
nanomole/Liter (nmol/L) | 11973.25 (NA) — Adjusted geometric standard error=1.07 | 11583.25 (NA) — Adjusted geometric standard error=1.07
Statistical Analysis 1: Comparison: Caffeine (Reference (R)) vs BI 730357 + Caffeine (Test (T)); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of GLSMs [%] = 96.74, 90% CI 2-sided [91.55 to 102.23] — Ratio of Geometric Least Squares Means (GLSMs) was calculated as (GLSM of "BI 730357 + caffeine"/GLSM of "caffeine"). Intra-individual geometric coefficient of variation (gCV [%]) = 8.6

3. Primary Outcome: Area Under the Concentration-time Curve of S-warfarin in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity, S-warfarin)
Description: Warfarin sodium is a racemic mixture of the R-and S-enantiomers. Area under the concentration-time curve of S-warfarin in plasma over the time interval from 0 extrapolated to infinity (AUC0-infinity,S-warfain) is reported.
Time Frame: Within 2 hours (h) predose for period 1, within 15 minutes predose for period 2 and 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 48 h, 71 h, 95 h, 119 h, 143 h after warfarin administration in both periods.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This set included all subjects in the TS who provided at least 1 PK endpoint that was defined as primary and was not excluded due to a clinical trial protocol (CTP) deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS, even if the subject contributed only 1 PK parameter value for 1 period to the statistical assessment.
Measure: Geometric Least Squares Mean (Standard Error); unit: hours * nanomole/Liter (h*nmol/L)
Groups:
- Warfarin (Reference (R)): In period 1 (Visit 2): Participants were administered 2 tablets of 5 milligram (mg) (total dose 10 mg) of warfarin sodium (Coumadin® 5 mg) orally as a single dose once on Day 1 of period 1 (Visit 2).
- BI 730357 + Warfarin (Test (T)): In period 2 (Visit 3): Participants were administered 3 film-coated tablets of 100 mg BI 730357 orally twice daily (bid) with daily dose 600 mg from Day -14 to Day 6 of Visit 3 (20 days in total). On the 15th day of BI 730357 treatment (Day 1 of Visit 3, 1 h after the morning dose of BI 730357), 2 tablets of 5 milligram (mg) (total dose 10 mg) of warfarin sodium (Coumadin® 5 mg) were administered orally once. The two warfarin sodium administrations were separated by a wash-out period of at least 20 days.
Arm/Group | Warfarin (Reference (R)) | BI 730357 + Warfarin (Test (T))
Number analyzed (Participants) | 16 | 16
hours * nanomole/Liter (h*nmol/L) | 55770.25 (NA) — Adjusted geometric standard error=1.10 | 61559.60 (NA) — Adjusted geometric standard error=1.10
Statistical Analysis 1: Comparison: Warfarin (Reference (R)) vs BI 730357 + Warfarin (Test (T)); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of GLSMs [%] = 110.38, 90% CI 2-sided [107.15 to 113.71] — Ratio of Geometric Least Squares Means (GLSMs) was calculated as (GLSM of "BI 730357 + warfarin"/GLSM of "Warfarin"). Intra-individual geometric coefficient of variation (gCV [%]) =4.8

4. Primary Outcome: Maximum Measured Concentration of the S-warfarin in Plasma (Cmax, S-warfarin)
Description: Warfarin sodium is a racemic mixture of the R-and S-enantiomers. Maximum measured concentration of the S-warfarin in plasma (Cmax) is reported.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/Liter (nmol/L)
Arm/Group | Warfarin (Reference (R)) | BI 730357 + Warfarin (Test (T))
Number analyzed (Participants) | 16 | 16
nanomole/Liter (nmol/L) | 1622.94 (NA) — Adjusted geometric standard error=1.05 | 1760.38 (NA) — Adjusted geometric standard error=1.05
Statistical Analysis 1: Comparison: Warfarin (Reference (R)) vs BI 730357 + Warfarin (Test (T)); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of GLSMs [%] = 108.47, 90% CI 2-sided [104.11 to 113.01] — Ratio of Geometric Least Squares Means (GLSMs) was calculated as (GLSM of "BI 730357 + warfarin"/GLSM of "Warfarin"). Intra-individual geometric coefficient of variation (gCV [%]) = 6.6

5. Primary Outcome: Area Under the Concentration-time Curve of Omeprazole in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity, Omeprazole)
Description: Area under the concentration-time curve of omeprazole in plasma over the time interval from 0 extrapolated to infinity (AUC0-infinity, omeprazole) is reported.
Time Frame: Within 2 hours (h) predose for period 1, within 15 minutes predose for period 2 and 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h after omeprazole administration in both periods.
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hours * nanomole/Liter (h*nmol/L)
Groups:
- Omeprazole (Reference (R)): In period 1 (Visit 2): Participants were administered 1 tablet of 20 mg of omeprazole (Antra MUPS® 20 mg gastro-resistant tablet) orally as a single dose once on Day 1 of period 1 (Visit 2).
- BI 730357 + Omeprazole (Test (T)): In period 2 (Visit 3): Participants were administered 3 film-coated tablets of 100 mg BI 730357 orally twice daily (bid) with daily dose 600 mg from Day -14 to Day 6 of Visit 3 (20 days in total). On the 15th day of BI 730357 treatment (Day 1 of Visit 3, 1 h after the morning dose of BI 730357), 1 tablet of 20 mg of omeprazole (Antra MUPS® 20 mg gastro-resistant tablet) was administered orally once. The two omeprazole administrations were separated by a wash-out period of at least 20 days.
Arm/Group | Omeprazole (Reference (R)) | BI 730357 + Omeprazole (Test (T))
Number analyzed (Participants) | 13 | 12
hours * nanomole/Liter (h*nmol/L) | 933.62 (NA) — Adjusted geometric standard error=1.22 | 931.22 (NA) — Adjusted geometric standard error=1.23
Statistical Analysis 1: Comparison: Omeprazole (Reference (R)) vs BI 730357 + Omeprazole (Test (T)); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of GLSM [%] = 99.74, 90% CI 2-sided [89.66 to 110.95] — Ratio of Geometric Least Squares Means (GLSM) was calculated as (GLSM of "BI 730357 + omeprazole"/GLSM of "Omeprazole"). Intra-individual geometric coefficient of variation (gCV [%]) =12.3

6. Primary Outcome: Maximum Measured Concentration of Omeprazole in Plasma (Cmax, Omeprazole)
Description: Maximum measured concentration of omeprazole in plasma (Cmax, omeprazole) is reported.
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/Liter (nmol/L)
Arm/Group | Omeprazole (Reference (R)) | BI 730357 + Omeprazole (Test (T))
Number analyzed (Participants) | 16 | 16
nanomole/Liter (nmol/L) | 504.07 (NA) — Adjusted geometric standard error=1.28 | 359.50 (NA) — Adjusted geometric standard error=1.28
Statistical Analysis 1: Comparison: Omeprazole (Reference (R)) vs BI 730357 + Omeprazole (Test (T)); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of GLSMs [%] = 71.32, 90% CI 2-sided [44.64 to 113.96] — Ratio of Geometric Least Squares Means (GLSMs) was calculated as (GLSM of "BI 730357 + omeprazole"/GLSM of "Omeprazole"). Intra-individual geometric coefficient of variation (gCV [%]) =87.8

7. Primary Outcome: Area Under the Concentration-time Curve of Midazolam in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity, Midazolam)
Description: Area under the concentration-time curve of midazolam in plasma over the time interval from 0 extrapolated to infinity (AUC0-infinity, midazolam) is reported.
Time Frame: Within 2 hours (h) predose for period 1, within 15 minutes predose for period 2 and 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h after midazolam administration in both periods.
Population: as for outcome 3
Measure: Geometric Least Squares Mean (Standard Error); unit: hours * nanomole/Liter (h*nmol/L)
Groups:
- Midazolam (Reference (R)): In period 1 (Visit 2): Participants were administered 1 milliliter (mL) oral solution of 2 mg of midazolam (Midazolam-ratiopharm® 2 mg/mL oral solution) orally as a single dose once on Day 1 of period 1 (Visit 2).
- BI 730357 + Midazolam (Test (T)): In period 2 (Visit 3): Participants were administered 3 film-coated tablets of 100 mg BI 730357 orally twice daily (bid) with daily dose 600 mg from Day -14 to Day 6 of Visit 3 (20 days in total). On the 15th day of BI 730357 treatment (Day 1 of Visit 3, 1 h after the morning dose of BI 730357), 1 milliliter (mL) oral solution of 2 mg of midazolam (Midazolam-ratiopharm® 2 mg/mL oral solution) was administered orally once. The two midazolam administrations were separated by a wash-out period of at least 20 days.
Arm/Group | Midazolam (Reference (R)) | BI 730357 + Midazolam (Test (T))
Number analyzed (Participants) | 16 | 16
hours * nanomole/Liter (h*nmol/L) | 56.81 (NA) — Adjusted geometric standard error=1.07 | 72.07 (NA) — Adjusted geometric standard error=1.07
Statistical Analysis 1: Comparison: Midazolam (Reference (R)) vs BI 730357 + Midazolam (Test (T)); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of GLSMs [%] = 126.85, 90% CI 2-sided [119.15 to 135.05] — Ratio of Geometric Least Squares Means (GLSMs) was calculated as (GLSM of "BI 730357 + midazolam"/GLSM of "Midazolam"). Intra-individual geometric coefficient of variation (gCV [%]) =10.1

8. Primary Outcome: Maximum Measured Concentration of Midazolam in Plasma (Cmax, Midazolam)
Description: Maximum measured concentration of midazolam in plasma (Cmax, midazolam) is reported.
Time Frame: as for outcome 7
Population: as for outcome 3
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/Liter (nmol/L)
Arm/Group | Midazolam (Reference (R)) | BI 730357 + Midazolam (Test (T))
Number analyzed (Participants) | 16 | 16
nanomole/Liter (nmol/L) | 19.09 (NA) — Adjusted geometric standard error=1.09 | 24.87 (NA) — Adjusted geometric standard error=1.09
Statistical Analysis 1: Comparison: Midazolam (Reference (R)) vs BI 730357 + Midazolam (Test (T)); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of GLSMs [%] = 130.25, 90% CI 2-sided [121.25 to 139.92] — Ratio of Geometric Least Squares Means (GLSMs) was calculated as (GLSM of "BI 730357 + midazolam"/GLSM of "Midazolam"). Intra-individual geometric coefficient of variation (gCV [%]) =11.6

ADVERSE EVENTS:
Time Frame: Cocktail: From 1st dose of cocktail until 1st dose of BI 730357 (BI) or end of 7 days residual effect period (REP) of cocktail, up to 7 days. BI: From 1st dose of BI until 2nd dose of cocktail, up to 14 days. BI+Cocktail: From 2nd dose of cocktail until last dose of BI+7 days of REP, up to 13 days. BI total: From 1st dose of BI until last dose of BI+7 days of REP, up to 27 days.
Description: Treated set (TS): The TS included all subjects who were entered and treated with at least 1 dose of trial drug.
Groups:
- Cocktail (Period 1): In period 1 participants were administered the cocktail reference treatment (R) consisting of 2 tablets of 50 milligrams (mg) (total dose 100 mg) of caffeine (Percoffedrinol® N 50 mg Tablets), 2 tablets of 5 mg (total dose 10 mg) of warfarin sodium (Coumadin® 5 mg), 1 tablet of 20 mg of omeprazole (Antra MUPS® 20 mg gastro-resistant tablet), and 1 milliliter (mL) oral solution of 2 mg of midazolam (Midazolam-ratiopharm® 2 mg/mL oral solution), each medication as a single dose, once on Day 1 of period 1 (Visit 2).
- BI 730357 (Period 2): In period 2 (Visit 3) participants were administered 3 film-coated tablets of 100 mg BI 730357 orally twice daily (bid) (daily dose 600 mg) from Day -14 until Day 1 of Visit 3, before the first dose of combination of BI and cocktail medications, (up to 14 days).
- BI 730357 + Cocktail (Period 2): In period 2 (Visit 3): Participants were administered 3 film-coated tablets of 100 mg BI 730357 orally twice daily (bid) (daily dose 600 mg) from Day 1 to Day 6 of Visit 3. On Day 1 of Visit 3, 1 h after the morning dose of BI 730357), the drug cocktail (100 mg caffeine, 10 mg warfarin, 20 mg omeprazole, and 2 mg midazolam) was administered orally once.
- BI 730357 Total: In period 2 (Visit 3): Participants were administered 3 film-coated tablets of 100 mg BI 730357 orally twice daily (bid) (daily dose 600 mg) from Day -14 to Day 6 of Visit 3 (20 days in total).
  The total number of adverse events due to BI 730357 in the second period is reported.
Arm/Group | Cocktail (Period 1) | BI 730357 (Period 2) | BI 730357 + Cocktail (Period 2) | BI 730357 Total
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 3/16 | 2/16 | 0/16 | 2/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cocktail (Period 1) (N=16) | BI 730357 (Period 2) (N=16) | BI 730357 + Cocktail (Period 2) (N=16) | BI 730357 Total (N=16)
Blepharospasm (Eye disorders) | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vessel puncture site haematoma (General disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT04679948/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT04679948/SAP_001.pdf